CLINICAL TRIAL: NCT01933880
Title: An Open, Self-Controlled, Prospective Study of Concerta on Cognitive Functions, Efficacy and Tolerance in the Pediatric Patients With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: A Long Term Post-Marketing Study on the EffIcacy and Safety of Osmotic Release Oral System (OROS) Methylphenidate on the Cognitive Functions of Attention Deficit Hyperactivity Disorder (ADHD) Participants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR016078; CONCERTAATT4099
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: Attention Deficit Hyperactivity Disorder; Methylphenidate Hydrochloride; CONCERTA
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OROS-MPH Group (Experimental): Participants with ADHD will receive OROS -MPH starting at initial dosage of 18 milligram per day (mg/d) which can be increased to 36 mg/d up to a maximum dosage of 54 mg/d according to the therapeutic effect and tolerance or maintained at 36 mg or re-adjusted to 18 mg due to intolerance.
  Interventions: Drug: Osmotic Release Oral System Methylphenidate Hydrochloride (OROS-MPH)
- Normal Group (Active Comparator): Participants did not receive any study drug in this group. Participants were assessed for changes in the cognitive functions and the efficacy was compared with ADHD children.
  Interventions: Other: No intervention

INTERVENTIONS:
Drug: Osmotic Release Oral System Methylphenidate Hydrochloride (OROS-MPH) — Osmotic release oral system methylphenidate hydrochloride (OROS-MPH) starting at initial dosage of 18 milligram per day (mg/d) which can be increased to 36mg/d up to a maximum dosage of 54mg/d according to the therapeutic effect and tolerance or maintained at 36 mg or re-adjusted to 18mg due to intolerance.
  Arms: OROS-MPH Group
Other: No intervention — Participants did not receive any study drug in this group. Participants were assessed for changes in the cognitive functions and the efficacy was compared with ADHD children.
  Arms: Normal Group

SUMMARY:
The purpose of this long term post-marketing study is to evaluate the effectiveness and safety of osmotic release oral system methylphenidate hydrochloride (OROS-MPH) in participants with Attention Deficit Hyperactivity Disorder (ADHD).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), prospective (study following participants forward in time), self-controlled, long-term post-marketing study in participants with ADHD. The study consists of 3 periods: screening period, wash-out period/run-in period (3 days), and open-label treatment period (12 weeks) which is divided into 2 periods that is dosage adjustment period and dose-optimization period. The total duration of the study is 12 weeks. During the dosage adjustment period, the dose of methylphenidate hydrochloride was adjusted to the optimal dose within 1-3 weeks starting with initial dosage of 18 milligram per day (mg/d) which can be increased to 36 mg/d up to a maximum dosage of 54 mg/d according to the therapeutic effect and tolerance or maintained at 36 mg or re-adjusted to 18 mg due to intolerance. Participants will receive the optimal dose determined during dose adjustment period for 9 weeks during the dose-optimization period. In the study, 2 types of participants will be enrolled in 2 groups (according to condition): OROS-MPH group (participants with ADHD) and the normal children group (healthy participants). The efficacy will be assessed primarily by Digit Span Test and Inattention /Over activity With Aggression (IOWA) Conners evaluation scale. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* ADHD children must sign the consent form in person, and their parents or guardian must endorse, in the consent form, participation of the child in the designated research program
* Through personal interaction and assessment questionnaire, examine to determine compliance of DSM-IV ADHD diagnostic criteria
* According to the judgment of researchers, the ADHD children should have normal intelligence. Normal intelligence is defined as no obvious evidence of mental retardation in general (specific learning disabilities will not be considered mental retardation in general), formal IQ test to be conducted and 85 marks or above ought to be scored
* ADHD children should not have been subjected to psychotropic drug treatment within 6 months. Those ADHD children on whom methylphenidate immediate-release tablets treatment is effective (with maximum daily dosage of 60 mg), may be admitted
* Normal children with IQ greater than or equal to 85

Exclusion Criteria:

* Unable to fully comply with the cognitive function test in the laboratory
* Known to be allergic to methylphenidate
* Consumption of psychoactive drugs currently or in the past 30 days, including use of monoamine oxidase inhibitors, clonidine, other alpha 2 adrenergic receptor agonists, tricyclic antidepressants, theophylline, bishydroxycoumarin etc
* History of alcohol, drugs or substances abuse
* Have medical history of type I or II bipolar affective disorder, anxiety disorder, schizophrenia or pervasive developmental disorder

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 194 (Actual)
Dates: Start 2009-12; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica Clinical trial, Study Director — Janssen Pharmaceutica
Locations (6):
- China (6):
  - Beijing
  - Changchun
  - Guangzhou
  - Hangzhou
  - Shanghai
  - Shenzhen

REFERENCES:
- [Derived] Zheng Y, Liang JM, Gao HY, Yang ZW, Jia FJ, Liang YZ, Fang F, Li R, Xie SN, Zhuo JM. An Open-label, Self-control, Prospective Study on Cognitive Function, Academic Performance, and Tolerability of Osmotic-release Oral System Methylphenidate in Children with Attention-deficit Hyperactivity Disorder. Chin Med J (Engl). 2015 Nov 20;128(22):2988-97. doi: 10.4103/0366-6999.168948. PMID 26608976

RESULTS

PARTICIPANT FLOW:
Groups:
- OROS-MPH Group: Participants with attention deficit hyperactivity disorder (ADHD) received osmotic release oral system-methylphenidate (OROS-MPH) tablets orally daily, starting at initial dosage of 18 milligram per day (mg/d) which could be increased to 36 mg/d up to a maximum dosage of 54 mg/d according to the therapeutic effect and tolerance or maintained at 36 mg or re-adjusted to 18 mg due to intolerance.
Period: Overall Study
Arm/Group | OROS-MPH Group | Normal Group
Started | 153 | 41
Completed | 123 | 40
Not Completed | 30 | 1
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Concomitant medication Interference | 0 | 1
Not completed — Followup exceeded 4 days to visit window | 19 | 0
Not completed — Other | 4 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) includes all of the subjects who received at least one study drug therapy and at least one efficacy evaluation. FAS for normal group included all participants who received baseline assessment scale evaluation and had at least one endpoint assessment scale evaluation.
Groups:
- Total: Total of all reporting groups
Arm/Group | OROS-MPH Group | Normal Group | Total
Number analyzed (Participants) | 128 | 40 | 168
Age, Customized [Number; unit: participants]
  Less than 7 to 8 Years | 48 (1.47) | 10 (1.72) | 58
  9 to 10 Years | 55 | 16 | 71
  11 to 12 Years | 25 | 14 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 108 | 23 | 131

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Digit Span Test Total Score at Week 12
Description: The digit span test is mainly used to measure the ability of short-term memory and attention. The participant will be given a string of digits and asked to repeat them forward, and then a second string of digits to repeat backward. The score is the number of correct responses, where the digits were repeated correctly. One point will be given for each correctly repeated string of digits. The maximum subscore in the Digits Forward is 16, and the maximum subscore in the Digits Backward is 14, summed for a total score of 30. A higher score is indicative of better recall and attention.
Time Frame: Baseline and Week 12
Population: Full Analysis Set (FAS) population for OROS-MPH Group included all participants who received at least one study drug therapy and had at least one efficacy evaluation. FAS for normal group included all participants who received baseline assessment scale evaluation and had at least one endpoint assessment scale evaluation.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 128 | 40
Scores on a scale
  Baseline | 11.7 (2.25) | 13.7 (2.43)
  Change at Week 12 | 1 (1.5) | 0.5 (1.48)
Statistical Analysis 1: Comparison: OROS-MPH Group; P-value was calculated to compare the data at Baseline and change at Week 12 for the OROS-MPH group; Test type: Superiority or Other; p = 0.0387, Signed Rank Sum Test

2. Primary Outcome: Change From Baseline in Inattention/Overactivity With Aggression (IOWA) Conners Behavior Rating Scale - I/O Score at Week 1
Description: IOWA Conners Behavior Rating Scale evaluated by parents provides accurate measurement standards for behavioral change and therapeutic response. It includes 2 sub-scales: Inattention/Overactivity (I/O) subscale and Attacks (A), also known as Opposition/Defiant (O/D) sub-scale. IO (primary measurement ) will be assessed using 5-items and all Items will be scored on a 4-point scale (from 0=not at all to 3=very much). Total score range is from 0 to 15. Higher scores indicate worsening.
Time Frame: Baseline and Week 1
Population: FAS population for OROS-MPH Group. Here "N" signifies number of participants who were evaluable for this outcome measure. Data for Normal group was not analyzed for IOWA Conners scale since as per the planned analysis normal participants were only analyzed for the memory effect in cognitive function test.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 127 | 0
Scores on a scale
  Baseline | 10 (2.4) |
  Change at Week 1 | -2.7 (2.18) |
Statistical Analysis 1: Comparison: OROS-MPH Group; P-value was calculated to compare the data at Baseline and change at Week 1 for the OROS-MPH group; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

3. Primary Outcome: Change From Baseline in IOWA Conners Behavior Rating Scale - I/O Score at Week 2
Description: as for outcome 2
Time Frame: Baseline and Week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 127 | 0
Scores on a scale
  Baseline | 10 (2.4) |
  Change at Week 2 | -4.1 (2.73) |
Statistical Analysis 1: Comparison: OROS-MPH Group; P-value was calculated to compare the data at Baseline and change at Week 2 for the OROS-MPH group; Test type: Superiority or Other; p = 0.0001, t-test, 2 sided

4. Primary Outcome: Change From Baseline in IOWA Conners Behavior Rating Scale - I/O Score at Week 3
Description: as for outcome 2
Time Frame: Baseline and Week 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 127 | 0
Scores on a scale
  Baseline | 10 (2.4) |
  Change at Week 3 | -5 (2.81) |
Statistical Analysis 1: Comparison: OROS-MPH Group; P-value was calculated to compare the data at Baseline and change at Week 3 for the OROS-MPH group; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

5. Primary Outcome: Change From Baseline in IOWA Conners Behavior Rating Scale - I/O Score at Week 7
Description: as for outcome 2
Time Frame: Baseline and Week 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 127 | 0
Scores on a scale
  Baseline | 10 (2.4) |
  Change at Week 7 | -5.8 (2.91) |
Statistical Analysis 1: Comparison: OROS-MPH Group; P-value was calculated to compare the data at Baseline and change at Week 7 for the OROS-MPH group; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

6. Primary Outcome: Change From Baseline in IOWA Conners Behavior Rating Scale - I/O Score at Week 12
Description: as for outcome 2
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 127 | 0
Scores on a scale
  Baseline | 10 (2.4) |
  Change at Week 12 | -6.2 (3.08) |
Statistical Analysis 1: Comparison: OROS-MPH Group; P-value was calculated to compare the data at Baseline and change at Week 12 for the OROS-MPH group; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

7. Secondary Outcome: Percentage of Participants With Total Score of IO Sub-scale Less Than or Equal to 5 in IOWA Conners Measurement Scale.
Description: Remission rate is the percentage of participants with total score of IO sub-scale less than or equal to 5 in IOWA Conners measurement scale
Time Frame: End of Week 1, 2, 3, 7 and 12
Population: FAS population for OROS-MPH Group included all participants who received at least one study drug therapy and had at least one efficacy evaluation. Data for Normal group was not analyzed for IOWA Conners scale since as per the planned analysis normal participants were only analyzed for the memory effect in cognitive function test.
Measure: Number; unit: Percentage of Participants
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 128 | 0
Percentage of Participants
  End of Week 1 | 25.98 |
  End of Week 2 | 51.97 |
  End of Week 3 | 66.93 |
  End of Week 7 | 78.74 |
  End of Week 12 | 81.10 |

8. Secondary Outcome: Stroop Color Word Naming Test
Description: This is a psychological test to observe the interference in which disparity between the meaning and color affects reading speed. A participant will be given 3 tasks of recognition: reading the printed colored ink (Color Test), reading color words in black ink (Word Test), and interference, reading color words printed in different colored ink (Word-Color Test). The test is scored on the number of correct answers. There are 100 items for each of the three categories and if they made it through the 100 words with time remaining, they would repeat the list. Median naming time in the Stroop color word naming test will be assessed. Stroop color word naming test 1 ,2 ,3 and 4 stand for gradually increased difficulty and each test has a corresponding baseline and endpoint.
Time Frame: Baseline and End of Week 12
Population: FAS for OROS-MPH Group included participants who took at least 1 study drug therapy and had at least 1 efficacy evaluation. FAS for normal group included participants who had baseline assessment scale evaluation and had at least 1 endpoint assessment scale evaluation. 'n'=participants who were evaluable at each specific time point for each arm.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 128 | 40
Seconds
  Test 1: Baseline (n=128, 40) | 20.561 (17.5433) | 6.213 (2.3174)
  Test 1: End of Week 12 (n=111, 40) | 18.961 (5.4474) | 5.7 (1.8355)
  Test 2: Baseline (n=128, 40) | 19.32 (14.8072) | 7.15 (2.6341)
  Test 2: End of Week 12 (n=111, 40) | 18.281 (13.6981) | 6.675 (2.2886)
  Test 3: Baseline (n=128, 40) | 18.652 (14.5219) | 6.875 (2.6451)
  Test 3: End of Week 12 (n=111, 40) | 16.946 (12.1586) | 6.513 (2.3898)
  Test 4: Baseline (n=128, 40) | 22.868 (11.3502) | 11.763 (4.4202)
  Test 4: End of Week 12 (n=111, 40) | 19.388 (9.8989) | 10.488 (4.2176)

9. Secondary Outcome: Wisconsin Card Sorting Test (WCST): Administered Responses (Ra) of Completed Examination
Description: WCST is used to evaluate participants' abilities of abstract generalization, working memory, and distraction-cognitive clinically, which reflects participants' cognitive function objectively and comprehensively. WCST consists of 13 test indicators and all indicators will be analyzed separately. The 13 indicators are as follows: number of trials administered; number of categories completed; response corrects; percent corrects; total number of errors; trials to complete first category; percent conceptual level responses; perseverative responses; perseverative errors; percent perseverative errors; nonperseverative errors; failure to maintain set; learning to learn. During number of trials administered or administered responses, participants were administered 128 cards and asked to sort the cards until all the 6 sorting categories was completed. Response number used to complete all 6 categories ranges from 50 to 128, lesser the better.
Time Frame: Baseline and End of Week 12
Population: FAS population for OROS-MPH Group included participants who received at least 1 study drug and had at least one efficacy evaluation. FAS for normal group included all participants who had baseline scale evaluation and had at least one endpoint scale evaluation. "n" signifies participants who were evaluable at each time point for each specific arm.
Measure: Mean (Standard Deviation); unit: Responses
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 128 | 40
Responses
  Baseline (n=128, 40) | 125.1 (8.74) | 120.8 (5.53)
  End of Week 12 (n=111, 40) | 116.4 (17.68) | 117.1 (17.37)

10. Secondary Outcome: WCST: Completed Categories (Cc)
Description: WCST is used to evaluate participants' abilities of abstract generalization, working memory, and distraction-cognitive clinically, which reflects participants' cognitive function objectively and comprehensively. WCST consists of 13 test indicators and all indicators will be analyzed separately. The 13 indicators are as follows: number of trials administered; number of categories completed; response corrects; percent corrects; total number of errors; trials to complete first category; percent conceptual level responses; perseverative responses; perseverative errors; percent perseverative errors; nonperseverative errors; failure to maintain set; learning to learn. In completed categoriies, number of categories completed out of 6 sorting categories after the test was evaluated. Ranges from 0 to 6. The more the number of categories completed the better is the response.
Time Frame: Baseline and End of Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Nunber of Categories Completed
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 128 | 40
Nunber of Categories Completed
  Baseline (n=128, 40) | 3.2 (1.56) | 3.3 (1.68)
  End of Week 12 (n=111, 40) | 4.1 (1.54) | 4 (1.34)

11. Secondary Outcome: WCST: Correct Responses (Rc)
Description: WCST is used to evaluate participants' abilities of abstract generalization, working memory, and distraction-cognitive clinically, which reflects participants' cognitive function objectively and comprehensively. WCST consists of 13 test indicators and all indicators will be analyzed separately. The 13 indicators are as follows: number of trials administered; number of categories completed; response corrects; percent corrects; total number of errors; trials to complete first category; percent conceptual level responses; perseverative responses; perseverative errors; percent perseverative errors; nonperseverative errors; failure to maintain set; learning to learn. The number of correct responses which meets all the requirements according to the response principles was evaluated. Ranges from 0-116, the more the better.
Time Frame: Baseline and End of Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: number of correct responses
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 128 | 40
number of correct responses
  Baseline (n=128, 40) | 72.9 (15.65) | 77.9 (12.27)
  End of Week 12 (n=111, 40) | 80.3 (12.25) | 84.7 (12.3)

12. Secondary Outcome: WCST: Error Responses (Re)
Description: WCST is used to evaluate participants' abilities of abstract generalization, working memory, and distraction-cognitive clinically, which reflects participants' cognitive function objectively and comprehensively. WCST consists of 13 test indicators and all indicators will be analyzed separately. The 13 indicators are as follows: number of trials administered; number of categories completed; response corrects; percent corrects; total number of errors; trials to complete first category; percent conceptual level responses; perseverative responses; perseverative errors; percent perseverative errors; nonperseverative errors; failure to maintain set; learning to learn. Number of error responses which did not comply with the response principles was evaluated. Ranges from 0 to 128, the less the better.
Time Frame: Baseline and End of Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: number of error responses
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 128 | 40
number of error responses
  Baseline (n=128, 40) | 52.3 (18.59) | 42.9 (17.77)
  End of Week 12 (n= 111, 40) | 36.1 (16.93) | 32.3 (15.11)

13. Secondary Outcome: WCST: Percentage of Correct Responses (Rc%)
Description: WCST is used to evaluate participants' abilities of abstract generalization, working memory, and distraction-cognitive clinically, which reflects participants' cognitive function objectively and comprehensively. WCST consists of 13 test indicators and all indicators will be analyzed separately. The 13 indicators are as follows: number of trials administered; number of categories completed; response corrects; percent corrects; total number of errors; trials to complete first category; percent conceptual level responses; perseverative responses; perseverative errors; percent perseverative errors; nonperseverative errors; failure to maintain set; learning to learn. Percentage of correct responses which meets all the requirements according to the response principles was evaluated. Ranges from 0 to 100 percent (%), the more the better.
Time Frame: Baseline and End of Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Percentage of correct responses
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 128 | 40
Percentage of correct responses
  Baseline (n=128, 40) | 58.678 (13.8072) | 65.52 (12.6227)
  End of Week 12 (n=111, 40) | 70.096 (11.6311) | 73.34 (10.5072)

14. Secondary Outcome: WCST: First Response (Rf)
Description: WCST is used to evaluate participants' abilities of abstract generalization, working memory, and distraction-cognitive clinically, which reflects participants' cognitive function objectively and comprehensively. WCST consists of 13 test indicators and all indicators will be analyzed separately. The 13 indicators are as follows: number of trials administered; number of categories completed; response corrects; percent corrects; total number of errors; trials to complete first category; percent conceptual level responses; perseverative responses; perseverative errors; percent perseverative errors; nonperseverative errors; failure to maintain set; learning to learn. Number of responses needed to complete the first color classification was evaluated. Ranges from 9 to 128, the lesser the better.
Time Frame: Baseline and End of Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: number of first responses
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 128 | 40
number of first responses
  Baseline (n=128,40) | 22.6 (22.29) | 25.2 (24.45)
  End of Week 12 (n=111, 40) | 23.4 (19) | 26.5 (22.77)

15. Secondary Outcome: WCST: Percentage of Conceptual Level Responses (Rf%)
Description: WCST is used to evaluate participants' abilities of abstract generalization, working memory, and distraction-cognitive clinically, which reflects participants' cognitive function objectively and comprehensively. WCST consists of 13 test indicators and all indicators will be analyzed separately. The 13 indicators are as follows: number of trials administered; number of categories completed; response corrects; percent corrects; total number of errors; trials to complete first category; percent conceptual level responses; perseverative responses; perseverative errors; percent perseverative errors; nonperseverative errors; failure to maintain set; learning to learn. Percentage of the responses completed with 3-10 continuous correct during the entire measuring process was evaluated. Ranges from 0 to 100%, the more the better.
Time Frame: Baseline and End of Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage of conceptual level responses
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 128 | 40
percentage of conceptual level responses
  Baseline (n=128, 40) | 46.36 (18.589) | 54.73 (18.48)
  End of Week 12 (n=111, 40) | 61.07 (17.244) | 65 (16.036)

16. Secondary Outcome: WCST: Perseverative Responses (Rp)
Description: WCST is used to evaluate participants' abilities of abstract generalization, working memory, and distraction-cognitive clinically, which reflects participants' cognitive function objectively and comprehensively. WCST consists of 13 test indicators and all indicators will be analyzed separately. The 13 indicators are as follows: number of trials administered; number of categories completed; response corrects; percent corrects; total number of errors; trials to complete first category; percent conceptual level responses; perseverative responses; perseverative errors; percent perseverative errors; nonperseverative errors; failure to maintain set; learning to learn. Number of perseverative responses were the responses which applied continuity principle for matching answers was evaluated. Ranges from 0 to 100, the less the better.
Time Frame: Baseline and End of Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: number of perseverative responses
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 128 | 40
number of perseverative responses
  Baseline (n=128, 40) | 33.7 (20.47) | 26.5 (14.09)
  End of Week 12 (n=111, 40) | 22 (16.21) | 18.6 (12.97)

17. Secondary Outcome: WCST: Perseverative Error Responses (Rpe)
Description: WCST is used to evaluate participants' abilities of abstract generalization, working memory, and distraction-cognitive clinically, which reflects participants' cognitive function objectively and comprehensively. WCST consists of 13 test indicators and all indicators will be analyzed separately. The 13 indicators are as follows: number of trials administered; number of categories completed; response corrects; percent corrects; total number of errors; trials to complete first category; percent conceptual level responses; perseverative responses; perseverative errors; percent perseverative errors; nonperseverative errors; failure to maintain set; learning to learn. Perseverative error responses are the number of responses which applied continuity principle for matching answers and also had the wrong answer was evaluated. Ranges from 0 to 128, the less the better.
Time Frame: Baseline and End of Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: number of perseverative error responses
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 128 | 40
number of perseverative error responses
  Baseline (n=128, 40) | 28.7 (15.24) | 23 (11.03)
  End of Week 12 (n=111, 40) | 19.4 (12.54) | 16.4 (9.85)

18. Secondary Outcome: WCST: Percentage of Perseverative Error Responses (Rpe%)
Description: WCST is used to evaluate participants' abilities of abstract generalization, working memory, and distraction-cognitive clinically, which reflects participants' cognitive function objectively and comprehensively. WCST consists of 13 test indicators and all indicators will be analyzed separately. The 13 indicators are as follows: number of trials administered; number of categories completed; response corrects; percent corrects; total number of errors; trials to complete first category; percent conceptual level responses; perseverative responses; perseverative errors; percent perseverative (pvt) errors; nonperseverative errors; failure to maintain set; learning to learn. Percentage of persistent errors out of total number of responses was evaluated. Ranges from 0 to 100%, the less the better.
Time Frame: Baseline and End of Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Percentage of pvt error responses
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 128 | 40
Percentage of pvt error responses
  Baseline (n=128, 40) | 22.67 (11.658) | 18.45 (8.083)
  End of Week 12 (n=111, 40) | 16.07 (9.188) | 13.59 (7.167)

19. Secondary Outcome: WCST: Non-Persistent Error Responses (nRpe)
Description: WCST is used to evaluate participants' abilities of abstract generalization, working memory, and distraction-cognitive clinically, which reflects participants' cognitive function objectively and comprehensively. WCST consists of 13 test indicators and all indicators will be analyzed separately. The 13 indicators are as follows: number of trials administered; number of categories completed; response corrects; percent corrects; total number of errors; trials to complete first category; percent conceptual level responses; perseverative responses; perseverative errors; percent perseverative errors; nonperseverative errors; failure to maintain set; learning to learn. Non perseverative error responses are the errors remaining after subtracting persistent errors from total errors. Ranges from 0 to 128 and was not linear (cannot be considered to be good or bad just judged by the number, analyzed with other factors case by case).
Time Frame: Baseline and End of Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: number of non-persistent error responses
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 128 | 40
number of non-persistent error responses
  Baseline (n=128, 40) | 23.54 (11.606) | 19.98 (8.94)
  End of Week 12 (n=111, 40) | 16.75 (9.241) | 15.8 (7.737)

20. Secondary Outcome: WCST: Failure to Maintain Set (Fm)
Description: WCST is used to evaluate participants' abilities of abstract generalization, working memory, and distraction-cognitive clinically, which reflects participants' cognitive function objectively and comprehensively. WCST consists of 13 test indicators and all indicators will be analyzed separately. The 13 indicators are as follows: number of trials administered; number of categories completed; response corrects; percent corrects; total number of errors; trials to complete first category; percent conceptual level responses; perseverative responses; perseverative errors; percent perseverative errors; nonperseverative errors; failure to maintain set; learning to learn. The frequency (number of times) of responses completed with 5 to 9 continuous correct was evaluated. Ranges from 0 to 26 and was not linear (cannot be considered to be good or bad just judged by the number, analyzed with other factors case by case).
Time Frame: Baseline and End of Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 128 | 40
number of times
  Baseline (n=128, 40) | 1.7 (1.62) | 2.3 (1.65)
  End of Week 12 (n=111, 40) | 2 (1.78) | 2.5 (1.75)

21. Secondary Outcome: WCST: Learning to Learn (L-C)
Description: WCST is used to evaluate participants' abilities of abstract generalization, working memory, and distraction-cognitive clinically, which reflects participants' cognitive function objectively and comprehensively. WCST consists of 13 test indicators and all indicators will be analyzed separately. "Learning to learn" indicator was a measure of decrement in the number of responses needed to achieve each successive category. The raw score ranged from 0 to 100. The high, negative value suggests the participants could not effectively learn the task presented by the WCST. Only calculated in those completed 3 or more categories and not linear (cannot be considered to be good or bad just judged by the number, analyzed with other factors case by case).
Time Frame: Baseline and End of Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: number of responses
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 128 | 40
number of responses
  Baseline (n=128, 40) | -2.49 (6.451) | -2.37 (6.31)
  End of Week 12 (n=111, 40) | -1.87 (3.85) | -1.34 (4.391)

22. Secondary Outcome: Coding Test
Description: The coding Test is a common test indicator for perceptual speed. The test presents a series of corresponding relationship between graphics and symbols to the participant, and then participants will be required to fill out the appropriate symbol following single symbol in the test part. The test is limited within 150 seconds and evaluated the number of symbols been replaced correctly by the participants.
Time Frame: Baseline and End of Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Number of symbols correctly replaced
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 128 | 40
Number of symbols correctly replaced
  Baseline (n=128, 40) | 63.4 (40.14) | 77.4 (44.83)
  End of Week 12 (n=111, 40) | 73.2 (41.41) | 83.1 (44.19)

23. Secondary Outcome: Academic Achievement
Description: Mathematics and language scores will be obtained from their corresponding examinations at school. Scores ranges from 0-100 respectively. Mathematics and language would be summarized separately.
Time Frame: Baseline and End of Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | OROS-MPH Group | Normal Group
Number analyzed (Participants) | 128 | 40
scores on a scale
  Chinese Achievement: Basline (n=128, 40) | 77.35 (13.791) | 94.21 (4.301)
  Chinese Achievement: End of Week 12(n=111, 40) | 83.94 (10.737) | 94.56 (4.396)
  Mathematical Achievement (MA):Baseline (n=128, 40) | 78.86 (15.407) | 96.23 (3.641)
  MA: End of Week 12 (n=111, 40) | 86.05 (11.579) | 96.13 (3.625)

24. Secondary Outcome: Number of Participants With Clinical Global Impression - CGI Scale Score
Description: CGI is an overall rating scale. Clinical Global Impression (Improvement of Diseases) is divided into seven grades: 1=very significant improvement, 24=significant improvement or advanced, 3=improvement or slightly advanced, 4=no change, 5=slight aggravation, 6=significant aggravation, and 7=very significant aggravation or seriously aggravated. Number of participants in each category of grade were assessed.
Time Frame: End of Week 1, 2, 3, 7 and 12
Population: as for outcome 7
Measure: Number; unit: Participants
Groups:
- Normal: Participants did not receive any study drug in this group. Participants were assessed for changes in the cognitive functions and the efficacy was compared with ADHD children.
Arm/Group | OROS-MPH Group | Normal
Number analyzed (Participants) | 128 | 0
Participants
  Significantly Advanced: End of Week 1 | 20 |
  Significantly Advanced: End of Week 2 | 28 |
  Significantly Advanced: End of Week 3 | 29 |
  Significantly Advanced: End of Week 7 | 35 |
  Significantly Advanced: End of Week 12 | 36 |
  Advanced: End of Week 1 | 59 |
  Advanced: End of Week 2 | 53 |
  Advanced: End of Week 3 | 44 |
  Advanced: End of Week 7 | 41 |
  Advanced: End of Week 12 | 46 |
  Slightly Advanced: End of Week 1 | 33 |
  Slightly Advanced: End of Week 2 | 28 |
  Slightly Advanced: End of Week 3 | 33 |
  Slightly Advanced: End of Week 7 | 28 |
  Slightly Advanced: End of Week 12 | 25 |
  No Change: End of Week 1 | 15 |
  No Change: End of Week 2 | 10 |
  No Change: End of Week 3 | 11 |
  No Change: End of Week 7 | 7 |
  No Change: End of Week 12 | 3 |
  Slightly Aggravated: End of Week 1 | 0 |
  Slightly Aggravated: End of Week 2 | 2 |
  Slightly Aggravated: End of Week 3 | 0 |
  Slightly Aggravated: End of Week 7 | 3 |
  Slightly Aggravated: End of Week 12 | 1 |
  Aggravated: End of Week 1 | 0 |
  Aggravated: End of Week 2 | 0 |
  Aggravated: End of Week 3 | 0 |
  Aggravated: End of Week 7 | 0 |
  Aggravated: End of Week 12 | 0 |
  Seriously Aggravated: End of Week 1 | 0 |
  Seriously Aggravated: End of Week 2 | 0 |
  Seriously Aggravated: End of Week 3 | 0 |
  Seriously Aggravated: End of Week 7 | 0 |
  Seriously Aggravated: End of Week 12 | 0 |

25. Secondary Outcome: Change From Baseline in I/O Score of IOWA Conners Behavior Rating Scale at Week 12
Description: IOWA conners behavior rating scale score in different dosage groups will be accessed to evaluate relationship between therapeutic effect and dosage. IOWA Conners Behavior Rating Scale evaluated by parents provides accurate measurement standards for behavioral change and therapeutic response. It includes 2 sub-scales: Inattention/Overactivity (I/O) subscale and Attacks (A), also known as Opposition/Defiant (O/D) sub-scale. IO (primary measurement ) will be assessed using 5-items and all Items will be scored on a 4-point scale (from 0=not at all to 3=very much). Total score range is from 0 to 15. Higher scores indicate worsening.
Time Frame: Baseline and End of Week 12
Population: FAS population for OROS-MPH Group included all participants who received at least one study drug therapy and had at least one efficacy evaluation. Here "N" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- OROS-MPH Group 18 Milligram (mg): Participants with ADHD received OROS -MPH tablets orally daily at a dose of 18 milligram per day (mg/d).
- OROS-MPH Group 36 mg: Participants with ADHD received OROS -MPH tablets orally daily at a dose of 36 milligram per day (mg/d)
- OROS-MPH Group 54 mg: Participants with ADHD received OROS -MPH tablets orally daily at a dose of 56 milligram per day (mg/d)
Arm/Group | OROS-MPH Group 18 Milligram (mg) | OROS-MPH Group 36 mg | OROS-MPH Group 54 mg
Number analyzed (Participants) | 86 | 30 | 1
Scores on a scale
  Baseline | 10 (2.42) | 10.3 (2.39) | 7 (0)
  Change at End of Week 12 | -6.8 (2.82) | -5.8 (3.32) | -4 (0)

26. Secondary Outcome: Change From Baseline in Total Scores of Digit Span Test at Week 12
Description: The digit span test total score will be accessed in different dosage groups to evaluate the relationship between therapeutic effect and dosage. The digit span test is mainly used to measure the ability of short-term memory and attention. The participant will be given a string of digits and asked to repeat them forward, and then a second string of digits to repeat backward. The score is the number of correct responses, where the digits were repeated correctly. One point will be given for each correctly repeated string of digits. The maximum subscore in the Digits Forward is16, and the maximum subscore in the Digits Backward is 14, for a total score of 30. A higher score was indicative of better recall and attention.
Time Frame: Baseline and End of Week 12
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | OROS-MPH Group 18 Milligram (mg) | OROS-MPH Group 36 mg | OROS-MPH Group 54 mg
Number analyzed (Participants) | 86 | 30 | 1
Scores on a scale
  Baseline | 11.7 (2.4) | 11.3 (1.95) | 15 (0)
  Change at End of Week 12 | 1.2 (1.54) | 0.8 (1.56) | 0 (0)

27. Secondary Outcome: Change From Baseline in Completion Time of Stroop Color-word Test at Week 12
Description: Completion time of stroop color-word test in different dosage groups will be accessed to evaluate the relationship between therapeutic effect and dosage. This is a psychological test to observe the interference in which disparity between the meaning and color affects reading speed. A participant will be given 3 tasks of recognition: reading the printed colored ink (Color Test), reading color words in black ink (Word Test), and interference, reading color words printed in different colored ink (Word-Color Test). The test will be scored on the number of correct answers. There are 100 items for each of the three categories and if they made it through the 100 words with time remaining, they would repeat the list. Median time of the naming time in the Stroop color word naming test will be accessed. Stroop color word naming test 1 ,2 ,3 and 4 stand for gradually increased difficulty and each test has a corresponding baseline and endpoint.
Time Frame: Baseline and End of Week 12
Population: FAS population for OROS-MPH Group included all participants who received at least one study drug therapy and had at least one efficacy evaluation. Here "N" signifies participants who were evaluable for this outcome measure and "n" signifies participants who were evaluable at each time point for each specific arm.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | OROS-MPH Group 18 Milligram (mg) | OROS-MPH Group 36 mg | OROS-MPH Group 54 mg
Number analyzed (Participants) | 86 | 30 | 1
Seconds
  Test 1: Baseline (n=86, 30, 1) | 22.229 (18.7304) | 17.7 (13.654) | 5 (0)
  Test 1: Change at End of Week 12 (n=82, 27, 1) | -3.318 (5.6413) | -1 (4.308) | 0 (0)
  Test 2: Baseline (n=86, 30, 1) | 20.538 (15.3567) | 17.29 (11.7025) | 9 (0)
  Test 2: Change at End of Week 12 (n=82, 27, 1) | -2.164 (5.2669) | -1.233 (3.9809) | 0 (0)
  Test 3: Baseline (n=86, 30, 1) | 19.515 (14.6203) | 17.473 (14.2673) | 7 (0)
  Test 3: Change at End of Week 12 (n=82, 27, 1) | -2.336 (5.3987) | -2.996 (6.6313) | 3 (0)
  Test 4: Baseline (n=86, 30, 1) | 23.61 (12.135) | 22.154 (9.2451) | 15 (0)
  Test 4: Change at End of Week 12 (n=82, 27, 1) | -4.374 (7.5921) | -3.974 (6.0143) | 1 (0)

28. Secondary Outcome: Percentage of Participants With Total Score of IO Sub-scale Less Than or Equal to 5 in IOWA Conners Measurement Scale at Week 12
Description: Remission rate in different dosage groups will be accessed to evaluate the relationship between therapeutic effect and dosage. Remission rate is the percentage of participants with total score of IO sub-scale less than or equal to 5 in IOWA Conners measurement scale.
Time Frame: Week 12
Population: as for outcome 25
Measure: Number; unit: Percentage of participants
Arm/Group | OROS-MPH Group 18 Milligram (mg) | OROS-MPH Group 36 mg | OROS-MPH Group 54 mg
Number analyzed (Participants) | 86 | 30 | 1
Percentage of participants | 85.37 | 74.07 | 100.00

29. Secondary Outcome: Number of Participants Compliant With Treatment
Description: Number of Participants who are Compliant with Treatment will be accessed. Less than 80 percent and more than 120 percent compliance signifies bad compliance, 80 to 120 percent compliance signifies good compliance . The compliance was calculated by the percentage of dose (actual dose multiplied by 100/theoretical dose).The theoretical dose means the dose prescribed by the Investigator.
Time Frame: End of Week 12
Population: FAS population for OROS-MPH Group. Here "N" signifies participants who were evaluable for this outcome measure. Data for Normal group was not analyzed for IOWA Conners scale since as per the planned analysis normal participants were only analyzed for the memory effect in cognitive function test.
Measure: Number; unit: participants
Arm/Group | OROS-MPH Group | Normal
Number analyzed (Participants) | 127 | 0
participants
  Less than 80 percent | 17 |
  Between 80 to 120 percent | 110 |
  More than 120 percent | 0 |

ADVERSE EVENTS:
Description: Safety Set for OROS-MPH Group included all participants who received at least one study drug therapy and at least one safety evaluation. Adverse events was not evaluated for normal group as participants did not receive any study drug in this group. Participants were only assessed for changes in the cognitive functions.
Arm/Group | OROS-MPH Group
Serious Adverse Events (participants affected / at risk) | 0/149
Other Adverse Events (participants affected / at risk) | 27/149
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OROS-MPH Group (N=149)
Loss of Appetite (Metabolism and nutrition disorders) | 19
Tinnitus (Ear and labyrinth disorders) | 1
Tonsillitis (Infections and infestations) | 1
Abnormal Heart Rate (Investigations) | 1
Decreased Blood Pressure (Investigations) | 2
Low sleep quality (Nervous system disorders) | 3
Headache (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 2
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Mouth and Pharynx Pain (Respiratory, thoracic and mediastinal disorders) | 1
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 3
Difficulty in falling asleep (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Irritability (Psychiatric disorders) | 1
Fever (General disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Difficulty in falling asleep (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days .In the event that issues arise regarding scientific integrity, the sponsor will review these issues with the investigator.